CLINICAL TRIAL: NCT04999774
Title: Análisis de la precisión de Ensayos de Laboratorio Para diagnóstico de Strongyloidiasis Humana en Escolares de Escuelas de áreas endémicas en Parroquias Del cantón San Lorenzo, Provincia de Esmeraldas, Ecuador
Brief Title: Evaluation of Strongyloidiasis in Ecuador: a fieLd Laboratory Accuracy Study
Acronym: ESTRELLA
Status: Completed | Type: Observational
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Collaborators: CECOMET (Centro de Epidemiologia Comunitaria y Medicina Tropical) (Unknown); Universidad Central del Ecuador (Other); World Health Organization (Other)
Responsible Party: Principal Investigator, Dora Buonfrate, Principal Investigator, IRCCS Sacro Cuore Don Calabria di Negrar
Other Study IDs: SCDonCalabria hospital
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Strongyloidiasis; Strongyloides Stercoralis Infection
MeSH Terms: conditions — Strongyloidiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- School-age children: Each SAC will be asked to supply fecal and blood samples for testing with:
  * Stool microscopy
  * Baermann method
  * Real-time PCR for S. stercoralis
  * Lateral flow rapid test
  * ELISA serology (NIE/SsIR and IgG Ratti)
  Interventions: Diagnostic Test: Different diagnostic tests

INTERVENTIONS:
Diagnostic Test: Different diagnostic tests — Each SAC will be tested with all tests
  Other Names: Baermann; Stool microscopy; Strongy Detect™ IgG ELISA Kit (InBios Manufacturer); Strongyloides Ratti IgG ELISA (Bordier Manufacturer); Real-time PCR; Lateral flow test

SUMMARY:
the World Health Organization (WHO) has recently committed to promote the control of strongyloidiasis within 2030 targets for STH control programmes. A specific target is to establish by 2030 an efficient strongyloidiasis control programme in school aged children (SAC), envisaging ivermectin preventive chemotherapy (PC) of SAC at risk of morbidity due to strongyloidiasis. The monitoring of such ambitious PC activity strictly requires appropriate diagnostic tools, but fundamental gaps exist in this field. Indeed, until now at the moment no consensus method for the diagnosis of S. stercoralis infection is recommended and the absence of a gold standard test limits capacity for effective diagnosis, surveillance and disease control. The aim of this project is to provide fundamental information on the performance and applicability of diagnostic methods for the assessment of S. stercoralis infection to inform the forthcoming WHO global strongyloidiasis control program to be implemented as a part of the WHO 2030 disease control targets. ESTRELLA is a cross-sectional study in an area of high prevalence of strongyloidiasis (San Lorenzo, Esmeraldas, Ecuador). The study will have a school-based approach, and each enrolled SAC will be asked to supply fecal and blood samples for testing with different methods for the diagnosis of S. stercoralis infection.

DETAILED DESCRIPTION:
Aim and objectives The aim of this project is to provide fundamental information on the performance and applicability of diagnostic methods for the assessment of S. stercoralis infection to inform the forthcoming WHO global strongyloidiasis control program to be implemented as a part of the WHO 2030 disease control targets.

Specific objectives are:

1. To estimate the accuracy of selected diagnostic methods currently available for the diagnosis of S. stercoralis;
2. To evaluate acceptability of each test and related sample collection method by the target population;
3. To assess the feasibility of each assay for the deployment as a field-based diagnostic, and as a monitoring and evaluation tool in endemic areas

Methods A cross-sectional study in an area of high prevalence of strongyloidiasis, based on previously-collected, preliminary data. The study will have a school-based approach.

Study area and participants The study will be conducted in Ecuador, in San Lorenzo, Esmeraldas province. Administratively, San Lorenzo is divided into 12 rural parishes (Alto Tambo, Ancón de Sardinas (Palma Real), Calderón, Carondelet, 5 de junio, Concepción, Mataje, San Javier de Cachavíì, Santa Rita, Tambillo, Tululbíì- Ricaurte, Urbina), two of which can only be reached by sea (Tambillo which is an island, and Ancon de Sardinas or Palma Real located on the shores of the ocean).

San Lorenzo health district has its headquarters in the capital city where there is a hospital with 75 beds and 4 basic specialties (medicine, paediatrics, gyneco-obstetrics and surgery), and a 24-hour health center for outpatient visits, laboratory tests, vaccinations, minor surgery and assistance with uncomplicated birth. In addition, there are 12 health centers in several localities, all recently renovated and equipped with electricity. In each health centre there is a team composed by a physician doctor, a nurse, a dentist, a midwife and a first-level health care worker. Health care is free, including medicines. However, supplies are often lacking. Community epidemiology activities and basic health care-training have been coordinated for years by the Cecomet team (Esmeraldas Center for Community Epidemiology and Tropical Medicine). Each health center covers variable number of villages, which receive a visit every 2/3 months from the health team. The latter carries out preventive activities, monitors chronic patients and specific groups at risk. Some health promoters, belonging to different ethnic groups, have been working on the territory for years as volunteers, with the role of community health supervisors and coordinators between teams and communities.

Every month, promoters and teams participate in a meeting coordinated by Cecomet with the aim to monitor the activities, discuss clinical cases and report the deaths. Participants are invited to discuss possible measures to prevent morbidity and mortality, and plan the next month's visits to the villages. The prevailing pathology reflects the epidemiological transition underway in many countries of the southern hemisphere: alongside the persistence of infectious / parasitic diseases such as malaria, Chagas disease, dengue, chikungunya, tuberculosis, and leishmaniasis, chronic degenerative pathology, especially hypertension and diabetes, has now considerable epidemiological importance. Intestinal parasites, given the scarcity or non-existence of basic services (safe water and sanitation) continues to be a major issue for children.

The study will take place in 5 of the 12 rural parishes of San Lorenzo, in the primary schools of 7 villages (Calderon, Carondelet, Ricaurte, S.Rita, S.Francisco del Bogotà, La Boca, Tambillo) mainly inhabited by Afro-descendants.

Study procedures Informative and educational meetings will be held in each community to inform the population about strongyloidiasis, the objectives of the study and the methodology for collecting samples. In this regard, educational leaflets, and audiovisual media adapted to the local population culture will be used.

Dates for intervention will be planned in agreement with the communities, the local authorities and the school managers. Informed consent from parents/guardians of the children will be sought before study implementation.

The day of the study, each participant will be invited to supply faeces and blood (from finger prick) samples for the testing procedures, and will be treated (as PC) with ivermectin 200 mcg/Kg single dose and albendazole 400 mg single dose according to the international standards and local protocols. A Case Report Form (CRF) will be used to collect information on relevant symptoms and other relevant characteristics concerning the levels of sanitation. Each CRF will be marked with an anonymized ID code, which will link the CRF to the samples supplied by each participant.

Faecal samples will be tested with Ritchie's formol-ether technique (for STH), Baermann method (specific for S. stercoralis), and with a real-time polymerase chain reaction (PCR) for S. stercoralis. For the latter test, part of the stool will be preserved in ethanol for transportation to the Laboratory of the Central University of Quito. Blood samples will be obtained by finger prick, and will be collected on filter papers for subsequent analysis with two ELISA assays (one based on crude antigen and one on a recombinant antigen) and a rapid dipstick test (RDT).

All tests will be carried out in the same country where samples are collected, in compliance with what required by a test to be used in control programmes.

Diagnostic tests

• Fecal tests Baermann method will be carried out according to the procedures described in the "Bench aids for the diagnosis of intestinal parasitosis", by the WHO.

The PCR is a real-time assay based on Verweji's method. Briefly, for DNA extraction, about 200 mg of feces are suspended in 200 µL of phosphate-buffered saline containing 2% polyvinylpolypyrolidone (Sigma-Aldrich) and frozen overnight at -20 °C until the extraction. After thawing and boiling, the samples are run by an automated extractor instrument (Magnapure LC.2, Roche). The real-time assay is performed as described previously. The amplification target is the small-subunit rRNA gene sequence for S. stercoralis. Appropriate positive and negative controls are included in all the experiments. As control for PCR inhibitors and amplification quality, the PhHV-1 control DNA is amplified with the appropriate primers/probe mix in the same reaction as S. stercoralis in multiplex PCR. The reactions, detection and data analysis are performed with the CFX96 detection system (Bio-Rad Laboratories). In a previous retrospective study the method demonstrated a sensitivity of 56.8% (95%CI 41.0-71.6)[10].

Serological tests

* The InBios Strongy Detect TM IgG ELISA detects specific IgG antibodies to Strongyloides recombinant antigens NIE and SsIR in serum. A previous kit included only NIE antigen, and the addition of SsIR aims at improving the performance of the test, which consists of an enzymatically amplified sandwich-type immunoassay. Positive and negative control samples are provided in the kit. The test will be run and interpreted according to the manufacturer's instruction.
* Bordier ELISA detects Strongyloides IgG antibodies by using somatic antigens from larvae of Strongyloides ratti. A previous retrospective study estimated its sensitivity and specificity at 90.8% (95%CI 85.8-95.7) and 94.0% (95%CI 91.2-96.9)[12], respectively. The test is performed as per manufacturer's instructions. However, as the cut-off varies between runs, we use a normalized Optical Density (OD) ratio to compare the results obtained in different sessions. A ratio ≥1 defines positive results. The test is widely available and deployed for routine screening and diagnostic activities across Europe.
* The RDT is a rapid dipstick test implemented by the Institute for Research in Molecular Medicine (INFORMM) of the University Sains Malaysia, Malaysia. A previous study reported sensitivity and specificity of 91.3% and 100%, respectively. The test result is qualitative, based on the appearance/absence of a colored test band 15 minutes after addition of the sample in the designated well. The presence of The test result two red colored lines (test and control lines) is interpreted as positive, whereas the dipstick that shows only one red line (control line) is interpreted as negative.

Sample size

For sample size calculation, sensitivity and specificity of the diagnostic tests to be evaluated were considered as follows:

TEST Sensitivity Specificity Baerman 0.5 0.98 ELISA Bordier 0.9 0.93

ELISA NIE 0.7 0.91

PCR 0.6 0.95

RDT 0.9 1.0

Sample size of 640 individuals was calculated for 95% confidence, 10% precision and an estimated prevalence of 15%.

Endpoints and Foreseen Analysis:

Demographic and clinical data will be summarized using descriptive statistics, measures of variability and precision and plots. Statistical tests will be used based on type of variables, tests assumptions and sample dimension. All parameters will be reported with 95% confidence intervals.

1. A) The sensitivity and specificity of the serologic assays and of the rapid test will be first calculated against the results of Baermann and PCR, both considered virtually 100% specific for the study purpose. Hence, the accuracy of each test will be calculated as the proportion of positive results over all positive (for sensitivity) and negative (for specificity) samples to Baermann and/or PCR. Uncertainty will be quantified by 95% confidence intervals.

   B) Considering that Baerman and PCR may have lower sensitivities than the other tests, which may result in misevaluation of (too low) specificity of the other tests, the sensitivity, specificity, negative predictive value (NPV) and positive predictive value (PPV) of all tests will be calculated also against a composite reference standard[16]. This will be based on a combination of the results of all tests, specifically: cases of strongyloidiasis will be identified as participants with positive PCR AND/OR Baermann AND/OR a positive serologic test plus the RDT OR two positive serologic tests. Moreover, in the latent class analysis (LCA) probabilistic models will be fitted in order to classify subjects as diseased or not diseased
2. The acceptability of the activity will be assessed as a) the number of people consenting to participate out of the whole target population to which participation to the study will be offered; b) the actual provision of the required faecal/blood samples by each consenting participant.
3. The feasibility of each technique will be evaluated a) calculating the number of samples for which a result of each technique will be available out of all suitable samples collected; when a result is not available, the reason (for instance problems with material transfer/ preservative/other technical reasons) will be collected b) investigating possible issues with a questionnaire administered to the laboratory personnel

ELIGIBILITY:
Inclusion Criteria:

* Children attending primary school in the selected communities

Exclusion Criteria:

* Refusal to participate
* Absence of written consent from parents/guardian

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: School age children attending the primary schools in the communities selected within the study area
Sampling Method: Non-Probability Sample
Enrollment: 781 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic test accuracy - primary reference standard | January-February 2022
  The sensitivity and specificity of the serologic assays and of the rapid test will be first calculated against the results of Baermann and PCR, both considered virtually 100% specific for the study purpose. Hence, the accuracy of each test will be calculated as the proportion of positive results over all positive (for sensitivity) and negative (for specificity) samples to Baermann and/or PCR. Uncertainty will be quantified by 95% confidence intervals.
Diagnostic test accuracy - composite reference standard | January-February 2022
  Considering that Baerman and PCR may have lower sensitivities than the other tests, which may result in misevaluation of (too low) specificity of the other tests, the sensitivity, specificity, negative predictive value (NPV) and positive predictive value (PPV) of all tests will be calculated also against a composite reference standard[16]. This will be based on a combination of the results of all tests, specifically: cases of strongyloidiasis will be identified as participants with positive PCR AND/OR Baermann AND/OR a positive serologic test plus the RDT OR two positive serologic tests. Moreover, in the latent class analysis (LCA) probabilistic models will be fitted in order to classify subjects as diseased or not diseased

SECONDARY OUTCOMES:
Acceptability | January 2022
  The acceptability of the activity will be assessed as a) the number of people consenting to participate out of the whole target population to which participation to the study will be offered; b) the actual provision of the required faecal/blood samples by each consenting participant.
Feasibility of in-field deployment of each test | January 2022
  The feasibility of each technique will be evaluated a) calculating the number of samples for which a result of each technique will be available out of all suitable samples collected; when a result is not available, the reason (for instance problems with material transfer/ preservative/other technical reasons) will be collected b) investigating possible issues with a questionnaire administered to the laboratory personnel

CONTACTS AND LOCATIONS:
Overall Officials: Angel Guevara, Principal Investigator — Universidad Central del Ecuador; Dora Buonfrate, Principal Investigator — IRCCS Sacro Cuore Don Calabria hospital
Locations (1):
- Centro de Epidemiologia Comunitaria y Medicina Tropical (CECOMET), Esmeraldas, Ecuador

IPD SHARING:
Plan to Share IPD: Yes
The dataset with raw anonymized data, will be either included in the pubblication or uploaded in an international datashering platform
Supporting Information: Study Protocol
Time Frame: After acceptance of pubblication of the main results of the study
Access Criteria: The dataset will be pubblicly available